CLINICAL TRIAL: NCT03445000
Title: A Single Arm Phase II Trial Evaluating the Activity of Alectinib for the Treatment of Pretreated RET-rearranged Advanced NSCLC
Brief Title: ALEctinib for the Treatment of Pretreated RET-rearranged Advanced Non-small Cell Lung Cancer
Acronym: ALERT-lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 12-17; 2017-002063-17 (EudraCT Number); MO30176 (Other: Roche)
Record Dates: First submitted 2018-01-05; First posted 2018-02-26 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer; Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Recurrent
Keywords: RET-rearrangement; advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial treatment (Experimental): Alectinib is administered orally, 600 mg, twice per day (1200 mg per day) until progression, refusal or unacceptable toxicity.
  Trial treatment may also continue beyond progression, with physician and patient agreement, for as long as the patient may still derive clinical benefit as per investigator decision.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Alectinib is administered orally 600mg (4x150mg capsules), twice per day (8 capsules, total 1200mg daily). The appropriate number of alectinib capsules will be provided to patients to be self-administered at home.
  Alectinib capsules must be taken at the same time each day with food. If a planned dose of alectinib is missed, patients can take the missed dose up until 6 hours before the next dose.
  Other Names: Alecensa

SUMMARY:
A research study to evaluate the activity of alectinib for the Treatment of pretreated patients with advanced NSCLC that have confirmed RETrearrangement.

DETAILED DESCRIPTION:
The trial is investigating the efficacy of alectinib in patients with advanced stage RET-rearranged NSCLC, treated with at least one platinum based systemic chemotherapy regimen. Preclinical studies have shown that alectinib, a highly selective next generation ALK inhibitor, has potent anti-tumour activity in RET-rearranged NSCLC. Therapeutically, several multiple kinases inhibitors, are potentially able to inhibit RET kinase function, which has been tested in several unselected NCSLC trials. However, those result were negative and none of the tested drugs was approved for lung cancer treatment.

The ALERT-lung trial is a single arm, phase II trial with the primary objective to assess the efficacy of alectinib in terms of best overall response (OR) assessed by RECIST v1.1 in selected NSCLC patients with RET rearrangement. The secondary objectives are to evaluate secondary measures of clinical efficacy including disease control, progression-free survival (PFS), and overall survival (OS) as well as to assess safety and tolerability of the treatment and to describe the association of primary and secondary outcomes with tumour characteristics.

Alectinib is administered orally, 600 mg, twice per day, until progression, refusal or unacceptable toxicity. Trial treatment may also continue beyond progression, with physician and patient agreement, for as long as the patient may still derive clinical benefit. A total sample size of 44 patients is required.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented non-small cell lung carcinoma
2. Advanced disease defined as recurrent stage IV (according to 8th TNM classification) or recurrent or progressive disease following multimodal therapy (radiation therapy, surgical resection, or definitive chemo-radiation therapy for locally advanced disease)
3. At least one prior platinum-based systemic regimen: Adjuvant or neoadjuvant or definitive platinum-based chemo-radiotherapy treatments are considered as a line of treatment only if completed less than 6 months before enrolment. Maintenance therapy following platinum doublet-based chemotherapy is not considered a separate regimen of therapy.
4. RET rearrangement detected by FISH, Nanostring or by parallel-sequencing on FFPE tumour tissue assessed locally.
5. Availability of FFPE tumour material for central confirmation of RETrearrangement
6. Measurable or non-measurable, but radiologically evaluable (except for skin lesions) disease according to RECIST v1.1 criteria
7. Age ≥18 years
8. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
9. Life expectancy >3 months
10. Adequate haematological function:

    * Haemoglobin ≥9 g/dL
    * Neutrophil count ≥1.5 ×109/L
    * Platelet count ≥100 × 109/L
    * WBC ≥2 ×109/L
11. Adequate renal function: Calculated creatinine clearance ≥45 mL/min (according to Cockcroft-Gault formula)
12. Adequate liver function:

    * Total bilirubin ≤2x ULN (except patients with Gilbert Syndrome, who can have total bilirubin ≤3.0 mg/dL)
    * ALT and AST ≤3x ULN (≤5x ULN for patients with concurrent liver ¨ metastasis)
13. Patient capable of proper therapeutic compliance, and accessible to correct followup.
14. Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine beta HCG pregnancy test within 7 days before enrolment into the trial and within 3 days before alectinib treatment start.
15. Sexually active men and women of childbearing potential must use an effective contraceptive method (intrauterine devices without hormones, bilateral tubal occlusion, vasectomized partner or total abstinence) during the trial treatment and for a period of at least 3 months following the last dose of alectinib.
16. Recovered from any previous therapy related toxicity to Grade ≤1 at date of enrolment (except for recovery to Grade ≤2 of alopecia, fatigue, creatinine increased, lack of appetite or peripheral neuropathy)
17. Written Informed Consent (IC) for trial treatment must be signed and dated by the patient and the investigator prior to any trial-related intervention.

Exclusion Criteria:

1. Untreated, active CNS metastases
2. Carcinomatous meningitis
3. Any previous (in the past 3 years) or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ ductal carcinoma of the breast
4. Any serious diseases or clinical conditions, including but not limited to uncontrolled active infection and any other serious underlying medical processes, that could affect the patient's capacity to participate in the trial
5. Liver disease characterized by:

   * ALT or AST >3 × ULN (>5 × ULN for patients with concurrent liver metastasis) confirmed on two consecutive measurements or
   * Impaired excretory function (e.g., hyperbilirubinaemia) or synthetic function or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminaemia, ascites, and bleeding from oesophageal varices or
   * Acute viral or active autoimmune, alcoholic, or other types of acute hepatitis
6. Patients with baseline symptomatic bradycardia
7. Previous treatment with any RET TKI or RET targeted therapy.
8. Known EGFR, ALK, ROS, and BRAF mutation (in addition to RET rearrangement)
9. Any concurrent systemic anticancer therapy.
10. Any GI disorder that may affect absorption of oral medications, such as malabsorption syndrome or status post major bowel resection.
11. History of hypersensitivity to any of the additives in the alectinib drug formulation.
12. Known HIV positivity or AIDS-related illness.
13. Women who are pregnant or in the period of lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enriqueta Felip, MD-PhD, Study Chair — Vall d'Hebron University Hospital; Jürgen Wolf, MD-PhD, Study Chair — University Hospital Cologne; Egbert F. Smith, MD-PhD, Study Chair — The Netherlands Cancer Institute Amsterdam
Locations (19):
- Institut Jules Bordet, Brussels, Belgium
- St. James Hospital, Dublin, Ireland
- Italy (4):
  - IRCCS Instituto Tumori Giovanni Paolo II, Bari
  - Instituto Europeo di Oncologia (IEO), Milan
  - University Hospital of Turin, Turin
  - Universita di Verona, Verona
- Netherlands (2):
  - The Netherlands Cancer Institute Amsterdam, Amsterdam
  - University Medical Center Maastricht, Maastricht
- Spain (8):
  - Hospital Teresa Herrara, A Coruña
  - Hospital general de Alicante, Alicante
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Quirón Dexeus, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
- Switzerland (3):
  - HFR Fribourg, Fribourg
  - Hôpital Universitaire de Genève, Geneva
  - UniversitatSpital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gainor JF, Shaw AT. Novel targets in non-small cell lung cancer: ROS1 and RET fusions. Oncologist. 2013;18(7):865-75. doi: 10.1634/theoncologist.2013-0095. Epub 2013 Jun 28. PMID 23814043
- [Result] Takeuchi K, Soda M, Togashi Y, Suzuki R, Sakata S, Hatano S, Asaka R, Hamanaka W, Ninomiya H, Uehara H, Lim Choi Y, Satoh Y, Okumura S, Nakagawa K, Mano H, Ishikawa Y. RET, ROS1 and ALK fusions in lung cancer. Nat Med. 2012 Feb 12;18(3):378-81. doi: 10.1038/nm.2658. PMID 22327623
- [Result] Lin JJ, Kennedy E, Sequist LV, Brastianos PK, Goodwin KE, Stevens S, Wanat AC, Stober LL, Digumarthy SR, Engelman JA, Shaw AT, Gainor JF. Clinical Activity of Alectinib in Advanced RET-Rearranged Non-Small Cell Lung Cancer. J Thorac Oncol. 2016 Nov;11(11):2027-2032. doi: 10.1016/j.jtho.2016.08.126. Epub 2016 Aug 17. PMID 27544060
- [Result] Gautschi O, Milia J, Filleron T, Wolf J, Carbone DP, Owen D, Camidge R, Narayanan V, Doebele RC, Besse B, Remon-Masip J, Janne PA, Awad MM, Peled N, Byoung CC, Karp DD, Van Den Heuvel M, Wakelee HA, Neal JW, Mok TSK, Yang JCH, Ou SI, Pall G, Froesch P, Zalcman G, Gandara DR, Riess JW, Velcheti V, Zeidler K, Diebold J, Fruh M, Michels S, Monnet I, Popat S, Rosell R, Karachaliou N, Rothschild SI, Shih JY, Warth A, Muley T, Cabillic F, Mazieres J, Drilon A. Targeting RET in Patients With RET-Rearranged Lung Cancers: Results From the Global, Multicenter RET Registry. J Clin Oncol. 2017 May 1;35(13):1403-1410. doi: 10.1200/JCO.2016.70.9352. Epub 2017 Mar 13. PMID 28447912
- [Result] Kodama T, Tsukaguchi T, Satoh Y, Yoshida M, Watanabe Y, Kondoh O, Sakamoto H. Alectinib shows potent antitumor activity against RET-rearranged non-small cell lung cancer. Mol Cancer Ther. 2014 Dec;13(12):2910-8. doi: 10.1158/1535-7163.MCT-14-0274. Epub 2014 Oct 27. PMID 25349307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period ranged from November 2018 to April 2020.
Pre-assignment Details: Overall, 15 patients were screened with 14 of them successfully enrolled in the trial (one patient was ineligible due to active CNS metastases).
Groups:
- Trial Treatment: Alectinib is administered orally, 600 mg, twice per day (1200 mg per day) until progression, refusal or unacceptable toxicity.
  Trial treatment may also continue beyond progression, with physician and patient agreement, for as long as the patient may still derive clinical benefit as per investigator decision.
  Alectinib: Alectinib is administered orally 600mg (4x150mg capsules), twice per day (8 capsules, total 1200mg daily). The appropriate number of alectinib capsules will be provided to patients to be self-administered at home.
  Alectinib capsules must be taken at the same time each day with food. If a planned dose of alectinib is missed, patients can take the missed dose up until 6 hours before the next dose.
Period: Overall Study
Arm/Group | Trial Treatment
Started | 14
Completed | 0 (Trial treatment is administered until progression, refusal or unacceptable toxicity.)
Not Completed | 14
Not completed — Disease progression | 8
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trial Treatment
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 60.6 [38.0 to 81.4]
Age, Customized [Count of Participants; unit: Participants]
  ≤ 60 years | 6
  >60 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 6
  Belgium | 1
  Italy | 2
  Spain | 5
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2: Ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours.
  Participants
    0 | 4
    1 | 10
Smoking status [Count of Participants; unit: Participants]
  Current | 1
  Former (≥ 100 cigarettes in the past during the whole life) | 3
  Never (0-99 cigarettes during the whole life) | 10

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR)
Description: Best overall response (OR = CR or PR), per investigator assessment. OR was determined using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). OR is defined as the best overall response [Complete Response (disappearance of all target and non-target lesions, no new lesions) or Partial Response (at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum of diameters, no measurable increase in a non-target lesion, no new lesions)] across all assessment points. Radiological tumour assessments were performed using CT scans.
Time Frame: Evaluated from enrollment through study completion, up to a maximum of 28 months.
Population: The efficacy cohort encompasses all evaluable patients, e.g. all enrolled patients excluding patients that were found to be ineligible (in retrospective review), patients that never started treatment and patients that were lost to follow-up before their first response evaluation (by RECIST 1.1). The efficacy cohort consists of 13 patients (there is one patient who was lost to follow-up before the first tumour assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Treatment
Number analyzed (Participants) | 13
Participants
  Complete response | 0
  Partial response | 0
  Stable disease | 9
  Non-Complete response/ Non-Progressive disease (in case of non-measurable disease only) | 1
  Progressive disease | 2
  Not evaluable | 1

2. Secondary Outcome: Disease Control at 24-weeks
Description: Best overall response of CR or PR, or SD (or non-CR/non-PD in the case of non-measurable disease only) by RECIST v1.1 criteria. Complete Response (CR): disappearance of all target and non-target lesions and no new lesions detected; Partial Response (PR): at least 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum of diameters (no measurable increase in a non-target lesion and no new lesion detected); Stable disease (SD): at most 20% increase or at most 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum of diameters (no measurable increase in a non-target lesion and no new lesion detected). Radiological tumour assessments were performed using CT scans.
Time Frame: From first documented response (CR, PR, SD, non-CR/non-PD) to 24 weeks or first documented progression or death from any cause, whichever came first, assessed every 8 weeks (±4 days).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Trial Treatment
Number analyzed (Participants) | 13
percentage of patients | 23.1 [5.0 to 53.8]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival time was measured from the date of enrolment until documented progression or death from any cause, whichever came first. PFS is assessed according to RECIST 1.1 criteria. Progressive disease: at least a 20% increase in the sum of the longest diameter of target lesions taking as reference the baseline sum of diameters, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Evaluated from enrollment through study completion, up to a maximum of 28 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trial Treatment
Number analyzed (Participants) | 13
months | 3.7 [1.8 to 7.3]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival time is measured from the date of enrolment until death from any cause.
Time Frame: Evaluated from enrollment through study completion, up to a maximum of 28 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trial Treatment
Number analyzed (Participants) | 13
months | NA [13.8 to NA] — Median survival time and upper limit are not determined as there was an insufficient number of participants with events.

5. Secondary Outcome: Number of Patients Experienced Adverse Events
Description: The safety and tolerability of alectinib treatment is assessed through analysis of the worst grade of toxicity/adverse events according to CTCAE v4.0 criteria observed over the whole treatment period.
Time Frame: Evaluated from enrollment through study completion, up to a maximum of 28 months.
Population: The safety cohort includes all patients who received at least one dose of trial treatment (i.e. all 14 patients).
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Treatment
Number analyzed (Participants) | 14
Participants
  Experienced adverse event(s) | 14
  Experienced serious adverse event(s) | 4

ADVERSE EVENTS:
Time Frame: Continuously from the date of Informed Consent signature until 30 days after all treatments discontinuation, up to approximately 28 months.
Description: Safety and tolerability of alectinib treatment is assessed through analysis of the worst grade of toxicity/adverse events according to CTCAE v4.0 criteria observed over the whole treatment period.
Arm/Group | Trial Treatment
All-Cause Mortality (participants affected / at risk) | 3/14
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trial Treatment (N=14)
Sudden death not otherwise specified (NOS) (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trial Treatment (N=14)
Fatigue (General disorders) | 6 (6)
Fever (General disorders) | 3 (3)
General disorders and administration site conditions - Other (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
CPK increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Olfactory nerve disorder (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03445000/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT03445000/SAP_001.pdf